CLINICAL TRIAL: NCT04599881
Title: A Phase 2 Open-Label Study of PTR-01 in Patients With Recessive Dystrophic Epidermolysis Bullosa (RDEB)
Brief Title: A Study of PTR-01 in Recessive Dystrophic Epidermolysis Bullosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phoenix Tissue Repair, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTR-01-002
Record Dates: First submitted 2020-10-08; First posted 2020-10-23 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
Keywords: RDEB
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Intervention Model Description: Open-label study
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PTR-01 3 mg/kg (Experimental): All patients will receive a PTR-01 dose of 3.0 mg/kg once weekly every week for a total of 4 doses, followed by a dose of 3.0 mg/kg every other week for a total of 7 doses.
  Interventions: Drug: PTR-01

INTERVENTIONS:
Drug: PTR-01 — IV recombinant collagen 7 at 3 mg/kg given weekly for 4 doses, followed by bi-weekly for 7 doses
  Other Names: Recombinant collagen 7; rC7

SUMMARY:
Protocol PTR-01-002 is a 3-part Phase 2, open-label study of PTR-01. While new patients will be enrolled, priority will be given to patients that satisfactorily completed study PTR-01-001.

DETAILED DESCRIPTION:
Protocol PTR-01-002 is a 3-part Phase 2, open-label study of PTR-01. While new patients will be enrolled, priority will be given to patients that satisfactorily completed study PTR-01-001.

In Part 1, patients will receive a dose of 3.0 mg/kg every week for a total of 4 doses. This will be followed by Part 2 in which patients will receive a dose of 3.0 mg/kg every other week for a total of 7 doses. In Part 3, patients will be followed for 12 weeks. No investigational therapy will be administered during this time. At the end of each dosing period, an efficacy assessment will be performed. Safety will be assessed continuously throughout the study.

Following the end of Part 3, patients may be eligible for a potential long-term extension to further refine the dosing regimen, depending upon study drug availability.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for study participation in the three month run in period of the study:

1. Willing to provide informed consent form, or if 12 to <18 years of age, legal guardian has provided informed consent form and the minor has signed an assent form acknowledging that they understand and agree to study procedures.
2. Has a diagnosis of RDEB based on genetic analysis and consistent with a recessive inheritance pattern.
3. Has deficient C7 staining at the dermal-epidermal junction (DEJ) by IF.
4. Agrees to use contraception as follows:

   For women of childbearing potential (WOCBP) agrees to use highly effective contraceptive (including abstinence) methods from Screening, through the study, and for at least 10 weeks after the last dose of study drug. Non-childbearing potential is defined as a female who meets either of the following criteria: age ≥50 years and no menses for at least 1 year or documented hysterectomy, bilateral tubal ligation, or bilateral oophorectomy.

   For males, agrees to use a condom with any WOCBP sexual partner from Day 1 of study treatment, through the study, and at least 10 weeks after the last dose of study drug.
5. Be willing and able to comply with this protocol.

Exclusion Criteria:

Patients with any of the following will be excluded from participation in the study:

1. Has known systemic hypersensitivity to any of the inactive ingredients in PTR-01.
2. Has previously had an anaphylactic reaction to PTR-01.
3. Is pregnant or nursing.
4. Has received in the last six months any investigational gene therapy product or in the last three months any non-gene therapy investigational products.
5. Is anticipated to receive new regimens of antibiotics or other anti-infectives during the trial.
6. Has any other medical or personal condition that, in the opinion of the Investigator, may potentially compromise the safety or compliance of the patient, or may preclude the patient's

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Wound healing | Up to 162 days
  Change in a majority of target lesions of at least 2 levels using a 7-point (1-7) Global Impression of Change instrument (7 being the worst)
Incidence of treatment-emergent adverse events | Up to 162 days
  Safety and tolerability, as assessed by treatment-emergent adverse events
Incidence of infusion-associated reactions | Up to 162 days
  Safety and tolerability, as assessed by infusion-associated reactions (IAR)
Incidence of anti-drug antibodies (ADA) | Up to 162 days
  Safety and tolerability, as assessed by immunogenicity through anti-drug antibody (ADA) testing

SECONDARY OUTCOMES:
Delivery of PTR-01 to skin | Up to 162 days
  PTR-01 incorporation by immunofluorescence using NC1 & NC2 staining, by dose frequency period
Formation of anchoring fibrils | Up to 162 days
  Formation of new anchoring fibrils as measured by electron microscopy
Change in wound surface area, as assessed by wound imaging | Up to 162 days
  Wound area of target lesions, as assessed by wound imaging
Change in wound surface area, as assessed by Investigator Global Impression of Change (IGIC) | Up to 162 days
  Wound area of target lesions, as assessed by IGIC
Change in total body wound surface area | Up to 162 days
  Change in total body wound surface area, using Rule of Nines
Change in skin integrity, as assessed by suction blister time | Up to 162 days
  Change in skin integrity, as assessed by suction blister time
Change in skin integrity, as assessed by time to re-blistering | Up to 162 days
  Change in skin integrity, as assessed by time to re-blistering
Change in itch severity, as assessed by modified Patient-Reported Outcome Measurement Information System (PROMIS) itch domains | Up to 162 days
  Severity of itch, as assessed by modified Patient-Reported Outcome Measurement Information System (PROMIS) itch domains
Change in itch severity, as assessed by the Instrument for Scoring Clinical Outcomes for Research of Epidermolysis Bullosa (iscorEB) | Up to 162 days
  Severity of itch, as assessed by Instrument for Scoring Clinical Outcomes for Research of Epidermolysis Bullosa (iscorEB), maximum score of 234 (worst)
Change in the impact of itch on quality of life | Up to 162 days
  Change in the impact of itch on quality of life, as assessed by the Pruritus-Specific Quality of Life Instrument (ItchyQoL), maximum score of 110 (worst)
Change in pain severity, as assessed by modified Patient-Reported Outcome Measurement Information System (PROMIS) pain domains | Up to 162 days
  Change in pain severity, as assessed by Patient-Reported Outcome Measurement Information System (PROMIS) pain domains
Change in pain severity, as assessed by the Instrument for Scoring Clinical Outcomes for Research of Epidermolysis Bullosa (iscorEB) | Up to 162 days
  Change in pain severity, as assessed by the Instrument for Scoring Clinical, maximum score of 234 (worst)
Change in the impact of pain on quality of life | Up to 162 days
  Change in the impact of pain on quality of life, as assessed by the Instrument for Scoring Clinical Outcomes for Research of Epidermolysis Bullosa (iscorEB) instrument, maximum score of 234 (worst)
Change of dysphagia, as assessed using the Brief Esophageal Dysphagia Questionnaire | Up to 162 days
  Change of dysphagia, as assessed using the Brief Esophageal Dysphagia Questionnaire, maximum score is 40 (worst)
Change in dysphagia, as assessed by volume of oral nutritional intake | Up to 162 days
  Change of dysphagia, as assessed by volume of oral nutritional intake, using patient interview and diary, maximum score is 40 (worst)
Stabilization of dysphagia, as assessed using the Brief Esophageal Dysphagia Scale | Up to 162 days
  Stabilization of dysphagia, as assessed using the Brief Esophageal Dysphagia Scale
Stabilization of dysphagia, as assessed by volume oral nutritional intake | Up to 162 days
  Stabilization of dysphagia, as assessed by volume oral nutritional intake, using patient interview and diary
Change in corneal symptoms | Up to 162 days
  Change of corneal symptoms (eye symptoms), as assessed by the Epidermolysis Bullosa Eye Disease Index (EB-EDI)
Stabilization of corneal symptoms | Up to 162 days
  Stabilization of corneal symptoms (eye symptoms), as assessed by the Epidermolysis Bullosa Eye Disease Index (EB-EDI)
Rate of change in nutritional markers (hemoglobin/hematocrit) | Up to 162 days
  Change of nutritional markers, as assessed by hemoglobin/hematocrit
Rate of change in nutritional markers (total protein/albumin) | Up to 162 days
  Change of nutritional markers, as assessed by total protein/albumin
Rate of change in nutritional markers (iron/TIBC) | Up to 162 days
  Change of nutritional markers, as assessed by iron/TIBC
Rate of change in nutritional markers (C-reactive protein) | Up to 162 days
  Change of nutritional markers, as assessed by C-reactive protein
Rate of stabilization of nutritional markers (hemoglobin/hematocrit) | Up to 162 days
  Stabilization of nutritional markers, as assessed by hemoglobin/hematocrit
Rate of stabilization of nutritional markers (total protein/albumin) | Up to 162 days
  Stabilization of nutritional markers, as assessed by total protein/albumin
Rate of stabilization of nutritional markers (iron/TIBC) | Up to 162 days
  Stabilization of nutritional markers, as assessed by iron/TIBC
Rate of stabilization of nutritional markers (C-reactive protein) | Up to 162 days
  Stabilization of nutritional markers, as assessed by C-reactive protein
Change in Investigator Global Impressions of Change (IGIC) | Up to 162 days
  Global impressions of change, as assessed through IGIC (1-7), 7 being worst
Change in Investigator Patient Impressions of Change (PGIC) | Up to 162 days
  Global impressions of change, as assessed through PGIC (1-7), 7 being worst
Change in disease activity and scarring | Up to 162 days
  Change in disease activity and scarring, as assessed by the Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI)
Change in overall quality of life, as assessed by the Quality of Life in Epidermolysis Bullosa (QOLEB) questionnaire | Up to 162 days
  Change in overall quality of life, as assessed by the Quality of Life in Epidermolysis Bullosa (QOLEB) questionnaire
Change in overall health | Up to 162 days
  Change in overall disability, as assessed by the Health Assessment Questionnaire or Children's Health Assessment Questionnaire (HAQ/CHAQ)
Change in mental health | Up to 162 days
  Change in mental health and social functioning, as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) mental health domains
Change in social function | Up to 162 days
  Change in mental health and social functioning, as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) social function domains
Change in amount of wound care | Up to 162 days
  Change in amount of wound care, as assessed by patient interviews
Change in time for wound care | Up to 162 daysUp to 162 days
  Change in time for wound care, as assessed by patient interviews
Change in cost of wound care | Up to 162 days
  Change in cost of wound care, as assessed by patient interviews
Change in overall patient impression of quality of life | Up to 162 days
  Change in overall quality of life, as assessed by patient interviews
Change in overall patient impression of disability | Up to 162 days
  Change in overall disability, as assessed by patient interviews

OTHER OUTCOMES:
Genotype/phenotype relationships | Up to 162 days
  Correlation between genotype (genetic mutation) and severity of disease
Impact of pharmacokinetics on safety outcomes | Up to 162 days
  Correlate Cmax and Area Under the Curve (AUC) with treatment emergent adverse events, infusion associated reactions and immune-mediated reactions
Impact of pharmacokinetics on efficacy outcomes | Up to 162 days
  Correlate Cmax and AUC with wound healing
Impact of pharmacokinetics on pharmacodynamic outcomes | Up to 162 days
  Correlate Cmax and AUC with suction blister time, C7 immunofluorescence on biopsy and formation of anchoring fibrils by electron microscopy

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Redwood City, California
  - Children's Hospital Colorado, Aurora, Colorado